CLINICAL TRIAL: NCT01045161
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Tolerability of 2 Doses of Aclidinium Bromide Compared With Placebo for 12 Weeks in Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease Followed by a 40-Week Evaluation of the Higher Aclidinium Bromide Dose
Brief Title: Efficacy, Safety, and Tolerability of Aclidinium Bromide in the Treatment of Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD) (LAS-MD-38)
Acronym: LAS-MD-38
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAS-MD-38
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Aclidinium bromide 200 μg dose twice per day, inhaled for 12 weeks of treatment At week 12, patients who were on Aclidinium bromide 200 μg will receive open label 400µg aclidinium bromide for 40 weeks
  Interventions: Drug: Aclidinium bromide
- 2 (Experimental): Aclidinium bromide 400 μg dose twice per day, inhaled for 12 weeks of treatment. At week 12, patients who were on Aclidinium bromide 400 μg will continue to receive open label 400µg aclidinium bromide for 40 weeks
  Interventions: Drug: Aclidinium bromide
- 3 (Placebo Comparator): Dose-match placebo, oral inhalation twice per day for 12 weeks of treatment. At week 12, patients who were on placebo will receive open label 400µg aclidinium bromide for 40 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide — Aclidinium bromide 200 μg, oral inhalation twice per day 12 weeks of treatment. At week 12, patients who were on Aclidinium bromide 200 μg will receive open label 400µg aclidinium bromide for 40 weeks of treatment.
  Arms: 1; 2
Drug: Placebo — Dose-matched placebo, oral inhalation twice per day for 12 weeks. At week 12, patients who were on placebo will receive open label 400 µg aclidinium bromide for 40 weeks of treatment
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of aclidinium bromide doses compared with placebo in the treatment of moderate to severe, stable chronic obstructive pulmonary disease. The study will be 56 weeks in duration; a 2-week run-in period followed by a 12-week double-blind, placebo-controlled treatment period. This will be followed by an open-label 40-week treatment period and a 2-week follow up phone call. All patients will receive the higher Aclidinium Bromide during the 40-week open label treatment period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stable moderate to severe COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, 2008; postbronchodilator FEV1/FVC < 70%, and postbronchodilator FEV1 ≥ 30% and < 80% predicted
* Current or former cigarette smokers

Exclusion Criteria:

* Patients who have been hospitalized for an acute COPD exacerbation within 3 months before the first visit
* Respiratory tract infection or COPD exacerbation in the 6 weeks before Visit 1
* Patient with any clinically significant respiratory conditions other than COPD, cardiovascular conditions or mental illness
* History or presence of asthma verified from medical records
* Chronic use of oxygen therapy greater than or equal to 15 hours per day
* Patient with uncontrolled infection due to HIV and/or active hepatitis
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics
* Patients with clinically significant cardiovascular conditions, including myocardial infarction during the previous 6 months, newly diagnosed arrhythmia within the previous 3 months, unstable angina, unstable arrhythmia that had required changes in pharmacological therapy or other intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, Ph. D., Study Director — AstraZeneca
Locations (112):
- United States (110):
  - Forest Investigative Site 1493, Birmingham, Alabama
  - Forest Investigative Site 1419, Birmingham, Alabama
  - Forest Investigative Site 1413, Muscle Shoals, Alabama
  - Forest Investigative Site 1353, Pell City, Alabama
  - Forest Investigative Site 1379, Phoenix, Arizona
  - Forest Investigative Site 2065, Fullerton, California
  - Forest Investigative Site 1451, National City, California
  - Forest Investigative Site 1388, Paramount, California
  - Forest Investigative Site 1424, Rolling Hill Estates, California
  - Forest Investigative Site 1427, Sacramento, California
  - Forest Investigative Site 1418, San Diego, California
  - Forest Investigative Site 2009, San Diego, California
  - Forest Investigative Site 1374, Torrance, California
  - Forest Investigative Site 1331, Vista, California
  - Forest Investigative Site 1380, Golden, Colorado
  - Forest Investigative Site 1447, Pueblo, Colorado
  - Forest Investigative Site 1364, Clearwater, Florida
  - Forest Investigative Site 1516, Edgewater, Florida
  - Forest Investigative Site 1403, Hollywood, Florida
  - Forest Investigative Site 1485, Homestead, Florida
  - Forest Investigative Site 1352, Miami, Florida
  - Forest Investigative Site 1391, Naples, Florida
  - Forest Investigative Site 1376, Port Orange, Florida
  - Forest Investigative Site 1372, South Miami, Florida
  - Forest Investigative Site 1407, Trinity, Florida
  - Forest Investigative Site 1185, Winter Park, Florida
  - Forest Investigative Site 1386, Atlanta, Georgia
  - Forest Investigative Site 1411, Calhoun, Georgia
  - Forest Investigative Site 1528, Lawrenceville, Georgia
  - Forest Investigative Site 0679, Coeur d'Alene, Idaho
  - Forest Investigative Site 1385, Elk Grove Village, Illinois
  - Forest Investigative Site 1409, O'Fallon, Illinois
  - Forest Investigative Site 1479, Anderson, Indiana
  - Forest Investigative Site 2022, Evansville, Indiana
  - Forest Investigative Site 1441, Indianapolis, Indiana
  - Forest Investigative Site 1149, South Bend, Indiana
  - Forest Investigative Site 1406, Iowa City, Iowa
  - Forest Investigative Site 1080, Topeka, Kansas
  - Forest Investigative Site 2033, Bowling Green, Kentucky
  - Forest Investigative Site 1090, Hazard, Kentucky
  - Forest Investigative Site 1430, New Orleans, Louisiana
  - Forest Investigative Site 1446, New Orleans, Louisiana
  - Forest Investigative Site 1360, Sunset, Louisiana
  - Forest Investigative Site 1412, Baltimore, Maryland
  - Forest Investigative Site 1518, North East, Maryland
  - Forest Investigative Site 1442, Brockton, Massachusetts
  - Forest Investigative Site 1421, Fall River, Massachusetts
  - Forest Investigative Site 1029, North Dartmouth, Massachusetts
  - Forest Investigative Site 1405, Chelsea, Michigan
  - Forest Investigative Site 0889, Livonia, Michigan
  - Forest Investigative Site 1487, Troy, Michigan
  - Forest Investigative Site 1128, Edina, Minnesota
  - Forest Investigative Site 1527, Fridley, Minnesota
  - Forest Investigative Site 1124, Minneapolis, Minnesota
  - Forest Investigative Site 1118, Rochester, Minnesota
  - Forest Investigative Site 1399, St Louis, Missouri
  - Forest Investigative Site 1400, Missoula, Montana
  - Forest Investigative Site 1354, Bellevue, Nebraska
  - Forest Investigative Site 1367, Bellevue, Nebraska
  - Forest Investigative Site 1476, Fremont, Nebraska
  - Forest Investigative Site 1363, Omaha, Nebraska
  - Forest Investigative Site 1390, Omaha, Nebraska
  - Forest Investigative Site 1422, Omaha, Nebraska
  - Forest Investigative Site 1359, Henderson, Nevada
  - Forest Investigative Site 1355, Las Vegas, Nevada
  - Forest Investigative Site 1486, Albuquerque, New Mexico
  - Forest Investigative Site 1489, Larchmont, New York
  - Forest Investigative Site 1425, New York, New York
  - Forest Investigative Site 1373, North Syracuse, New York
  - Forest Investigative Site 1392, Charlotte, North Carolina
  - Forest Investigative Site 1366, High Point, North Carolina
  - Forest Investigative Site 1136, Cincinnati, Ohio
  - Forest Investigative Site 1371, Cincinnati, Ohio
  - Forest Investigative Site 1361, Columbus, Ohio
  - Forest Investigative Site 1433, Columbus, Ohio
  - Forest Investigative Site 1530, Toledo, Ohio
  - Forest Investigative Site 1393, Zanesville, Ohio
  - Forest Investigative Site 1362, Oklahoma City, Oklahoma
  - Forest Investigative Site 2018, Medford, Oregon
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1377, Collegeville, Pennsylvania
  - Forest Investigative Site 1423, Erie, Pennsylvania
  - Forest Investigative Site 1428, Feasterville, Pennsylvania
  - Forest Investigative Site 1443, Philadelphia, Pennsylvania
  - Forest Investigative Site 1510, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1449, Tipton, Pennsylvania
  - Forest Investigative Site 1445, Johnston, Rhode Island
  - Forest Investigative Site 1477, Lincoln, Rhode Island
  - Forest Investigative Site 1144, Columbia, South Carolina
  - Forest Investigative Site 1517, Easley, South Carolina
  - Forest Investigative Site 1506, Grenville, South Carolina
  - Forest Investigative Site 1450, Union, South Carolina
  - Forest Investigative Site 1526, Fayetteville, Tennessee
  - Forest Investigative Site 1356, Knoxville, Tennessee
  - Forest Investigative Site 1417, Knoxville, Tennessee
  - Forest Investigative Site 1389, Amarillo, Texas
  - Forest Investigative Site 1440, Arlington, Texas
  - Forest Investigative Site 1494, Austin, Texas
  - Forest Investigative Site 1375, Houston, Texas
  - Forest Investigative Site 1444, Houston, Texas
  - Forest Investigative Site 1401, Houston, Texas
  - Forest Investigative Site 1381, Houston, Texas
  - Forest Investigative Site 1357, Hurst, Texas
  - Forest Investigative Site 1426, Plano, Texas
  - Forest Investigative Site 1410, Tomball, Texas
  - Forest Investigative Site 1480, Abingdon, Virginia
  - Forest Investigative Site 1402, Lynchburg, Virginia
  - Forest Investigative Site 1404, Norfolk, Virginia
  - Forest Investigative Site 1358, Richmond, Virginia
  - Forest Investigative Site 0988, Tacoma, Washington
- Canada (2):
  - Forest Investigative Site 1177, Vancouver, British Columbia
  - Forest Investigative Site 0969, Windsor, Ontario

REFERENCES:
- [Derived] Rennard SI, Scanlon PD, Ferguson GT, Rekeda L, Maurer BT, Garcia Gil E, Caracta CF. ACCORD COPD II: a randomized clinical trial to evaluate the 12-week efficacy and safety of twice-daily aclidinium bromide in chronic obstructive pulmonary disease patients. Clin Drug Investig. 2013 Dec;33(12):893-904. doi: 10.1007/s40261-013-0138-1. PMID 24085591
- See also: las-md-38-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4070&filename=las-md-38-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from December of 2009 to June of 2010 at 112 study sites (110 in the United States and 2 additional sites in Canada).
Pre-assignment Details: A total of 544 patients were randomized, with 542 in the Part A Safety population. Of the 454 patients who completed Part A, 448 patients continued into Part B, receiving at least 1 dose of open-label treatment, were included in the Part B Safety Population. Of these patients, 405 had a baseline and postbaseline assessment for the ITT Population.
Groups:
- Placebo - Part A Placebo to Aclidinium Bromide 400 μg - Part B: Dose matched placebo, twice per day, oral inhalation for 12 weeks of double-blind treatment. After 12 weeks, patients who were on placebo received open-label Aclidinium Bromide, 400 microgram dose, for an additional 40 weeks.
- Aclidinium Bromide 200μg to Aclidinium Bromide 400μg: Aclidinium bromide 200 microgram dose, oral inhalation, twice per day for 12 weeks of double-blind treatment. After 12 weeks, patients who were Aclidinium bromide 200 microgram dose, received open-label Aclidinium Bromide, 400 microgram dose, for an additional 40 weeks.
- Aclidinium Bromide 400μg to Aclidinium Bromide 400μg: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 12 weeks of double-blind treatment. After 12 weeks, patients continued to receive Aclidinium bromide, 400 microgram dose as an open-label treatment for an additional 40 weeks
Period: Part A - 12 Weeks Double Blind Treatment
Arm/Group | Placebo - Part A Placebo to Aclidinium Bromide 400 μg - Part B | Aclidinium Bromide 200μg to Aclidinium Bromide 400μg | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg
Started | 182 | 184 | 178
Completed | 151 | 155 | 148
Not Completed | 31 | 29 | 30
Not completed — Withdrawal by Subject | 8 | 12 | 6
Not completed — Adverse Event | 4 | 3 | 8
Not completed — Lack of Efficacy | 6 | 3 | 2
Not completed — COPD Exacerbation | 4 | 1 | 6
Not completed — Other Reason | 3 | 3 | 3
Not completed — Protocol Violation | 3 | 4 | 3
Not completed — Lost to Follow-up | 3 | 3 | 2
Period: Part B - 40 Additional Weeks Open Label
Arm/Group | Placebo - Part A Placebo to Aclidinium Bromide 400 μg - Part B | Aclidinium Bromide 200μg to Aclidinium Bromide 400μg | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg
Started | 147 | 154 | 147
Completed | 111 | 118 | 115
Not Completed | 36 | 36 | 32
Not completed — Withdrawal by Subject | 10 | 7 | 9
Not completed — Adverse Event | 10 | 10 | 7
Not completed — Lack of Efficacy | 3 | 5 | 5
Not completed — COPD Exacerbation | 1 | 5 | 1
Not completed — Other Reason | 4 | 2 | 1
Not completed — Protocol Violation | 3 | 6 | 3
Not completed — Lost to Follow-up | 5 | 1 | 6

BASELINE CHARACTERISTICS:
Population: A total of 544 patients were randomized, with 542 in the Part A Safety population. Of the 454 patients who completed Part A, 448 patients continued into Part B, receiving at least 1 dose of open-label treatment, were included in the Part B Safety Population. Baseline characteristics for Part B are based on participant totals of 147, 154 and 147
Groups:
- Placebo Part A / Placebo to Aclidinium Bromide 400μg Part B: Dose-matched placebo, twice per day, oral inhalation for 12 weeks of double-blind treatment in Part A of the Trial.
  After week 12 (conclusion of Part A), patients who were on placebo received open-label Aclidinium Bromide, 400 microgram dose, for an additional 40 weeks.
- Aclidinium Bromide(AB) 200μg Part A / AB 200μg to 400μg Part B: Aclidinium bromide 200 microgram dose, oral inhalation, twice per day for 12 weeks of double-blind treatment in Part A of the Trial.
  After week 12 (conclusion of Part A), patients who were on a double-blind, 200 microgram Aclidinium Bromide dose, were switched to open-label Aclidinium Bromide at a 400 microgram dose for an additional 40 weeks.
- Aclidinium Bromide(AB) 400μg Part A / AB 400μg to 400μg Part B: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 12 weeks of double-blind treatment in Part A of the Trial.
  After week 12 (conclusion of Part A), patients who were on a double-blind, 400 microgram Aclidinium Bromide dose, were switched to open-label Aclidinium Bromide at the same 400 microgram dose for an additional 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Part A / Placebo to Aclidinium Bromide 400μg Part B | Aclidinium Bromide(AB) 200μg Part A / AB 200μg to 400μg Part B | Aclidinium Bromide(AB) 400μg Part A / AB 400μg to 400μg Part B | Total
Number analyzed (Participants) | 182 | 183 | 177 | 542
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part A | 61.7 (9.3) | 63.4 (8.5) | 63.2 (9.0) | 62.8 (8.9)
  Part B | 61.3 (9.1) | 63.8 (8.2) | 63.1 (8.6) | 62.8 (8.7)
Age, Customized [Number; unit: participants]
  ≥ 40 to < 60 years - Part A | 72 | 57 | 57 | 186
  ≥ 60 to < 70 years - Part A | 72 | 79 | 77 | 228
  ≥ 70 years - Part A | 38 | 47 | 43 | 128
  ≥ 40 to < 60 years - Part B | 60 | 46 | 46 | 152
  ≥ 60 to < 70 years - Part B | 58 | 67 | 67 | 192
  ≥ 70 years - Part B | 29 | 41 | 34 | 104
Gender [Count of Participants; unit: Participants] — Part A
  Participants
    Female | 82 | 84 | 88 | 254
    Male | 100 | 99 | 89 | 288
Gender [Count of Participants; unit: Participants] — Part B
  Participants
    Female | 82 | 84 | 88 | 254
    Male | 100 | 99 | 89 | 288
Region of Enrollment [Number; unit: participants] — Part A
  participants
    United States | 180 | 181 | 175 | 536
    Canada | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants] — Part B
  participants
    United States | 145 | 152 | 145 | 442
    Canada | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part A: Morning Predose (Trough) Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from baseline in Trough forced expiratory volume in 1 second before the morning dose of aclidinium bromide, Last Observation Carried Forward (LOCF)
Time Frame: Change from baseline (Week 0) to Week 12
Population: Of 544 patients randomized, 542 patients received at least 1 dose of double-blind treatment and were included in the Safety Population. Of these patients, 541 had a baseline and at least 1 postbaseline FEV1 assessment and qualified for the Intent to Treat (ITT) Population.
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo: Dose-matched placebo twice per day, inhaled for 12 weeks of treatment.
- Aclidinium Bromide 200 μg: Aclidinium bromide 200 μg dose twice per day, inhaled for 12 weeks of treatment.
- Aclidinium Bromide 400 μg: Inhaled Aclidinium bromide 400 μg twice per day for 12 weeks.
Arm/Group | Placebo | Aclidinium Bromide 200 μg | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 182 | 182 | 177
L | -0.008 (0.015) | 0.043 (0.015) | 0.064 (0.016)
Statistical Analysis 1: Comparison: Placebo vs Aclidinium Bromide 200 μg; Test type: Superiority or Other; p = 0.019, ANCOVA; Least Squares Mean Difference = 0.051, 95% CI 2-sided [0.01 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs Aclidinium Bromide 400 μg; Test type: Superiority or Other; p = 0.0012, ANCOVA; Least squares mean difference = 0.072, 95% CI 2-sided [0.03 to 0.12]

2. Secondary Outcome: Part A: Peak Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from baseline in peak FEV1 at week 12, Last Observation Carried Forward (LOCF)
Time Frame: Change from baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | Placebo | Aclidinium Bromide 200 μg | Aclidinium Bromide 400 μg
Number analyzed (Participants) | 182 | 182 | 177
L | 0.087 (0.018) | 0.202 (0.018) | 0.212 (0.018)

3. Primary Outcome: Part B: Morning Predose (Trough) FEV1
Description: Change from Baseline in Morning Pre-dose (trough) Forced Expiratory Volume in 1 Second (FEV1) at Week 52, Lost Observation Carried Forward (LOCF)
Time Frame: Change from baseline (Week 0) to 52 Weeks
Population: A total of 544 patients were randomized, with 542 in the Part A Safety population. Of the 454 patients who completed Part A, 448 patients continued into Part B, receiving at least 1 dose of open-label treatment, were included in the Part B Safety Population. Of these patients, 405 had a baseline and postbaseline assessment for the ITT Population.
Measure: Mean (Standard Deviation); unit: L
Groups:
- Placebo - Aclidinium Bromide 400 μg: Dose matched placebo, oral inhalation, twice per day for 12 weeks of treatment. At week 12, patients who were on placebo were switched to open label 400µg aclidinium bromide for 40 weeks
- Aclidinium Bromide 200 μg - Aclidinium Bromide 400 μg: Aclidinium bromide, 200 μg dose, oral inhalation, twice per day for 12 weeks of treatment. At week 12, patients who were on Aclidinium bromide 200 μg were switched to open label 400µg aclidinium bromide for 40 weeks.
- Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg: Aclidinium bromide, 400 μg dose, oral inhalation, twice per day for 12 weeks of treatment. At week 12, patients received open label 400µg aclidinium bromide for 40 additional weeks
Arm/Group | Placebo - Aclidinium Bromide 400 μg | Aclidinium Bromide 200 μg - Aclidinium Bromide 400 μg | Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg
Number analyzed (Participants) | 134 | 139 | 132
L | 0.045 (0.021) | 0.029 (0.020) | 0.048 (0.021)
Statistical Analysis 1: Comparison: Placebo - Aclidinium Bromide 400 μg vs Aclidinium Bromide 200 μg - Aclidinium Bromide 400 μg; Test type: Superiority or Other; p = 0.0192, ANCOVA; Least Squares Mean Difference = 0.051, 95% CI 2-sided [0.01 to 0.09]
Statistical Analysis 2: Comparison: Placebo - Aclidinium Bromide 400 μg vs Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg; Test type: Superiority or Other; p = 0.0012, ANCOVA; Least Squares Mean difference = 0.072, 95% CI 2-sided [0.03 to 0.12]

4. Secondary Outcome: Part B: Peak FEV1
Description: Change from Baseline in Peak FEV1 (L) at Week 52, Last Observation Carried Forward (LOCF)
Time Frame: Change from baseline (Week 0) to 52 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo - Aclidinium Bromide 400 μg: Dose matched placebo, oral inhalation twice per day for 12 weeks. At week 12, patients who were on placebo switched to open label 400µg aclidinium bromide for 40 weeks
- Aclidinium Bromide 200 μg - Aclidinium Bromide 400 μg: Aclidinium bromide 200 μg, oral inhalation twice per day for 12 weeks of treatment. At week 12, patients who were on Aclidinium bromide 200 μg switched to open label 400µg aclidinium bromide for 40 weeks
- Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg: Aclidinium bromide 400 μg dose, oral inhalation twice per day for 12 weeks of treatment. At week 12, patients who were on Aclidinium bromide 400 μg switched to open label 400µg aclidinium bromide for 40 weeks
Arm/Group | Placebo - Aclidinium Bromide 400 μg | Aclidinium Bromide 200 μg - Aclidinium Bromide 400 μg | Aclidinium Bromide 400 μg - Aclidinium Bromide 400 μg
Number analyzed (Participants) | 134 | 139 | 132
L | 0.185 (0.023) | 0.176 (0.023) | 0.172 (0.023)

ADVERSE EVENTS:
Time Frame: Adverse Event reporting began in December of 2009 and concluded in July of 2011 at 112 study sites (110 in the United States and 2 additional sites in Canada).
Groups:
- Placebo - Part A: Dose matched placebo, twice per day, oral inhalation for 12 weeks of double-blind treatment.
- Aclidinium Bromide 200 μg - Part A: Aclidinium bromide 200 microgram dose, oral inhalation, twice per day for 12 weeks of double-blind treatment.
- Aclidinium Bromide 400 μg - Part A: Aclidinium bromide, 400 microgram dose, oral inhalation twice per day for 12 weeks of double-blind treatment.
- Placebo to Aclidinium Bromide 400 μg - Part B: After week 12 (conclusion of Part A), patients who were on placebo received open-label Aclidinium Bromide, 400 microgram dose, for an additional 40 weeks.
- Aclidinium Bromide 200μg to Aclidinium Bromide 400μg - Part B: Part B - After week 12 (conclusion of Part A), patients who were on a double-blind, 200 microgram Aclidinium Bromide dose, were switched to open-label Aclidinium Bromide at a 400 microgram dose for an additional 40 weeks.
- Aclidinium Bromide 400μg to Aclidinium Bromide 400μg - Part B: After week 12 (conclusion of Part A), patients who were on a double-blind, 400 microgram Aclidinium Bromide dose, were switched to open-label Aclidinium Bromide at the same 400 microgram dose for an additional 40 weeks.
Arm/Group | Placebo - Part A | Aclidinium Bromide 200 μg - Part A | Aclidinium Bromide 400 μg - Part A | Placebo to Aclidinium Bromide 400 μg - Part B | Aclidinium Bromide 200μg to Aclidinium Bromide 400μg - Part B | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg - Part B
Serious Adverse Events (participants affected / at risk) | 12/182 | 11/183 | 8/177 | 15/147 | 20/154 | 14/147
Other Adverse Events (participants affected / at risk) | 22/182 | 20/183 | 28/177 | 37/147 | 50/154 | 52/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part A (N=182) | Aclidinium Bromide 200 μg - Part A (N=183) | Aclidinium Bromide 400 μg - Part A (N=177) | Placebo to Aclidinium Bromide 400 μg - Part B (N=147) | Aclidinium Bromide 200μg to Aclidinium Bromide 400μg - Part B (N=154) | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg - Part B (N=147)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 5 | 4 | 7 | 3
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrenteritis salmonella (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonas bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Agitated depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Labyrinthitis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part A (N=182) | Aclidinium Bromide 200 μg - Part A (N=183) | Aclidinium Bromide 400 μg - Part A (N=177) | Placebo to Aclidinium Bromide 400 μg - Part B (N=147) | Aclidinium Bromide 200μg to Aclidinium Bromide 400μg - Part B (N=154) | Aclidinium Bromide 400μg to Aclidinium Bromide 400μg - Part B (N=147)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 21 | 16 | 23 | 24 | 35 | 41
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 3 | 9 | 9 | 8
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 6 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.